CLINICAL TRIAL: NCT02571049
Title: Randomized, Double-Blind, Crossover, Comparator Pilot Study of DFN-11 Injection (Strength A vs. Strength B) for Rapidly Escalating Migraine
Brief Title: Pilot Study of Two Different Strengths of DFN-11 Injection for Rapidly Escalating Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DFN-11-CD-006
Record Dates: First submitted 2015-10-01; First posted 2015-10-08 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-02

CONDITIONS: Rapidly Escalating Migraine
MeSH Terms: interventions — Sumatriptan

STUDY DESIGN:
Intervention Model Description: DFN-11 injection and placebo injection administered in one treatment period and two DFN-11 injections administered in another treatment period
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sumatriptan 3 mg then 6 mg (Experimental): DFN-11 (sumatriptan, 3 mg) and placebo first then two DFN-11 injections
  Interventions: Drug: DFN-11
- Sumatriptan 6 mg then 3 mg (Experimental): Two DFN-11 (sumatriptan, 3 mg) injections first then DFN-11 injection and placebo
  Interventions: Drug: DFN-11

INTERVENTIONS:
Drug: DFN-11 — Sumatriptan 3 mg versus 6 mg
  Other Names: Sumatriptan succinate injection

SUMMARY:
Pilot study to compare the efficacy and safety of two strengths of injections of subcutaneous DFN-11 in subjects with rapidly escalating migraine headaches.

DETAILED DESCRIPTION:
Pilot study to compare the proportion of subjects experiencing pain freedom at 60 minutes post-treatment between headache treated with Strength A of DFN-11 and Strength B of DFN-11

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of episodic migraine, with or without aura for at least 1 year prior to screening
2. Experience an average of 2 to 8 migraines per month for the past 12 months of which approximately 75% or more rapidly escalate to moderate or severe pain within 2 hours of onset
3. Females must:

   * be practicing an effective method of birth control (e.g. prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [e.g., condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel], or male partner sterilization) before entry and throughout the study, or
   * be surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), or
   * be postmenopausal (spontaneous amenorrhea for at least 1 year)
4. Females of child-bearing potential must have a negative urine pregnancy test at screening
5. Able and willing to read and comprehend written instructions and complete the electronic diary information required by the protocol
6. Must have internet access to complete daily headache diary

Exclusion Criteria:

1. Inability to distinguish migraine from other primary headaches
2. Experiences headache of any kind at a frequency greater than or equal to 15 days per month
3. Chronic opioid therapy (> 10 days in the 30 days prior to screening)
4. Current treatment with monoamine oxidase A (MAO-A) inhibitors or use within 4 weeks before randomization
5. Hemiplegic or basilar migraine
6. History, symptoms or signs of ischemic cardiac, cerebrovascular or peripheral vascular syndromes
7. Uncontrolled hypertension (screening systolic/diastolic blood pressure > 140/90 mmHg in 2 out of 3 readings)
8. History of epilepsy or conditions associated, which in the opinion of the Investigator, increase the likelihood of present day seizure
9. History (within 2 years) of drug or alcohol abuse as defined by DSM-IV-TR criteria.
10. Systemic disease, which in the opinion of the Investigator, would contraindicate participation
11. History of a neurological or psychiatric condition, which in the opinion of the Investigator would contraindicate participation
12. Pregnant or lactating women
13. Have taken any investigational medication within 30 days before randomization, or are scheduled to receive an investigational drug
14. Subjects with a positive urine drug screen for recreational drugs or marijuana (whether legal or not) or for prescription drugs not explained by stated concomitant medications
15. Clinical laboratory or electrocardiogram (ECG) abnormality that in the opinion of the Investigator would endanger the subject or interfere with the study conduct. If the results of the clinical laboratory or ECG are outside of normal reference range the subject may still be enrolled but only if these findings are determined to be not clinically significant by the Investigator. This determination must be recorded in the subject's source document prior to enrolment.
16. Fridericia's corrected QT (QTcF) interval greater than 450 msec
17. Severe renal impairment (creatinine > 2 mg/dl)
18. Serum total bilirubin > 2.0 mg/dL
19. Serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase > 2.5 times the upper limit of normal
20. Subjects who in the opinion of the investigator experience rebound headache from caffeine usage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinvest, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cady RK, Munjal S, Cady RJ, Manley HR, Brand-Schieber E. Randomized, double-blind, crossover study comparing DFN-11 injection (3 mg subcutaneous sumatriptan) with 6 mg subcutaneous sumatriptan for the treatment of rapidly-escalating attacks of episodic migraine. J Headache Pain. 2017 Dec;18(1):17. doi: 10.1186/s10194-016-0717-7. Epub 2017 Feb 7. PMID 28176235

RESULTS

PARTICIPANT FLOW:
Groups:
- Sumatriptan 3 mg Then 6 mg: Subjects were first dispensed one sumatriptan 3 mg autoinjector and one matching placebo autoinjector to self-administer consecutively in one migraine attack (total 3 mg active sumatriptan) and in the next study visit were dispensed two sumatriptan 3 mg autoinjectors to self-administer consecutively in another migraine attack (total 6 mg active sumatriptan).
- Sumatriptan 6 mg Then 3 mg: Subjects were first dispensed two sumatriptan 3 mg autoinjectors to self-administer consecutively in one migraine attack (total 6 mg active sumatriptan) and in the next study visit were dispensed one sumatriptan 3 mg autoinjector and one matching placebo autoinjector to self-administer consecutively in one migraine attack (total 3 mg active sumatriptan) .
Period: Screening
Arm/Group | Sumatriptan 3 mg Then 6 mg | Sumatriptan 6 mg Then 3 mg
Started | 10 | 14
Completed | 8 | 12
Not Completed | 2 | 2
Not completed — Did not meet entry criteria | 2 | 2
Period: Randomization
Arm/Group | Sumatriptan 3 mg Then 6 mg | Sumatriptan 6 mg Then 3 mg
Started | 8 | 12
Completed | 8 | 10
Not Completed | 0 | 2
Not completed — No migraine attack | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects who were randomized into the study
Arm/Group | All Subjects
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.80 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Reporting Pain Freedom at 60 Minutes Post-treatment
Time Frame: 60 minutes post-treatment
Measure: Number; unit: Percentage of responders
Groups:
- Sumatriptan 3 mg: DFN-11 active injection and placebo injection
- Sumatriptan 6 mg: Two DFN-11 active injections
Arm/Group | Sumatriptan 3 mg | Sumatriptan 6 mg
Number analyzed (Participants) | 18 | 19
Percentage of responders | 50 | 52.63

ADVERSE EVENTS:
Groups:
- Sumatriptan 3 mg SC: All subjects who had an AE when treated with sumatriptan 3 mg SC
- Sumatriptan 6 mg SC: All subjects who had an AE when treated with sumatriptan 6 mg SC
Arm/Group | Sumatriptan 3 mg SC | Sumatriptan 6 mg SC
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 14/20 | 18/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sumatriptan 3 mg SC (N=20) | Sumatriptan 6 mg SC (N=20)
Paraesthesia (Nervous system disorders) | 5 (5) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Flushing (General disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 0 (0) | 2 (2)
Muscle Contraction (General disorders) | 1 (1) | 2 (2)
Myalgia (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Hyperhidrosis (General disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Disorientation (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No